CLINICAL TRIAL: NCT06417073
Title: Effects of Task-Oriented Station Training on Cognitive and Hand Functions in Nursing Home Elders: Comparing Tele-Rehabilitation, Face-to-Face, and Home-Based Interventions
Brief Title: Effects of Task-Oriented Station Training on Cognitive Levels and Hand Functions in Geriatric Residents of Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Ceyhun Türkmen, Assoc. Prof., Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: d897232bb89442f7
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Decline; Motor Function Disorders; Geriatric Health
Keywords: Task-Oriented Station Training; Cognitive Function; Hand Function; Tele-Rehabilitation; Face-to-Face Intervention
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-to-Face Interventions (Experimental)
  Interventions: Behavioral: Face-To-Face Task-orianted Training
- Tele-Rehabilitation (Experimental)
  Interventions: Behavioral: Tele-Rehabilitation Task-orianted Training
- Home-Based Training (Experimental)
  Interventions: Behavioral: Home-based Task-orianted Training

INTERVENTIONS:
Behavioral: Face-To-Face Task-orianted Training — In this study, face-to-face task-oriented station training is provided by trained occupational therapists to elderly nursing home residents. Each session involves structured activities that simulate real-world challenges designed to improve cognitive and hand functions. These include exercises to enhance fine motor skills, hand strength, coordination, and cognitive tasks such as problem-solving and memory exercises.
  Arms: Face-to-Face Interventions
Behavioral: Tele-Rehabilitation Task-orianted Training — This intervention utilizes video-conferencing technology to deliver task-oriented training to elderly nursing home residents, focusing on cognitive and hand function improvements.
  Arms: Tele-Rehabilitation
Behavioral: Home-based Task-orianted Training — Home-Based Task-Oriented Training Intervention Description:
  This home-based intervention involves a series of task-oriented activities specifically designed to improve cognitive and hand functions for elderly residents in nursing homes. Participants carry out prescribed activities independently, based on detailed guides provided by occupational therapists. The activities are tailored to stimulate cognitive processes and enhance fine motor skills, including tasks like sorting, assembling, and manipulative exercises that replicate daily challenges. Each participant follows a structured program of daily 45-minute sessions for two weeks, with periodic remote check-ins by therapists to assess progress and adjust the difficulty of tasks as needed. This format allows participants to engage in rehabilitation at their own pace, within the comfort of their own living spaces, fostering greater autonomy and adherence to the intervention.
  Arms: Home-Based Training

SUMMARY:
This study explores the impact of task-oriented station training on the cognitive levels and hand functions of elderly residents in nursing homes. Utilizing methods like tele-rehabilitation, face-to-face sessions, and home-based programs, this research aims to determine the most effective approach for improving the cognitive and manual skills of this population. The hypothesis driving this study is that targeted task-oriented training can significantly improve the cognitive functions and hand dexterity of elderly individuals living in nursing homes, potentially enhancing their quality of life and independence. Participants receive different types of interventions-tele-rehabilitation, direct face-to-face training, and guided home programs-to evaluate which modality most effectively supports cognitive and hand function improvements. The study's design is randomized and assesses the outcomes through various established psychological and physical tests. With an aging global population, such strategies are crucial for maintaining the independence and quality of life of our elderly, potentially reducing the need for intensive care solutions and allowing for longer periods of self-sufficiency and well-being. This summary presents the study in a straightforward manner, explaining the purpose, hypothesis, methods, and significance of the research to make it accessible to non-specialist readers.

ELIGIBILITY:
**Inclusion Criteria:**

* Age 65 years and older.
* Residency in a nursing home.
* Able to provide informed consent, either directly or through a legal guardian.
* Sufficient cognitive function to participate in the intervention, as indicated by a Mini-Mental State Examination (MMSE) score of 18 or higher.
* Physically able to participate in task-oriented activities, with or without assistive devices.
* Stable medical condition, with no hospitalizations due to acute illness in the last three months prior to the study commencement.

**Exclusion Criteria:**

* Diagnosed with severe dementia or any cognitive impairment severe enough as per the healthcare provider to interfere with participation in the study.
* Any medical condition that significantly limits physical activity or requires intensive medical care during the study period, such as unstable cardiovascular disease, severe osteoarthritis, or recent fractures.
* Participation in any other experimental rehabilitation or drug trials concurrently.
* Severe sensory deficits that would prevent participation in the tasks (e.g., severe vision or hearing loss not correctable with aids).
* Life expectancy less than 6 months as estimated by a physician.
* Significant psychiatric disorders that might impair the ability to comply with study protocols.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function Using the Mini-Mental State Examination (MMSE) | Baseline (start of intervention), Post-intervention (immediately after the 2-week intervention),
  The Mini-Mental State Examination (MMSE) is a widely used tool for assessing cognitive function, which measures various aspects of cognitive abilities including orientation to time and place, immediate recall, short-term memory, language use, comprehension, and basic motor skills. The score ranges from 0 to 30, with higher scores indicating better cognitive function. This test will be used to quantify changes in cognitive levels of participants after undergoing task-oriented station training.

SECONDARY OUTCOMES:
Improvement in Hand Function Using the Nine-Hole Peg Test | Baseline and Post-intervention (immediately after the 2-week intervention).
  The Nine-Hole Peg Test measures dexterity and hand function. Participants are timed on how quickly they can place and then remove nine pegs into a pegboard with one hand. This test is used to evaluate fine motor skills improvement, particularly the ability to coordinate visually guided fine movements.
Quality of Life Changes Measured by the Short Form Health Survey (SF-36) | Baseline and Post-intervention (immediately after the 2-week intervention).
  The SF-36 is a survey used to assess quality of life across eight domains: physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality (energy/fatigue), social functioning, role limitations due to emotional problems, and mental health (psychological distress and psychological well-being). This measure will evaluate the impact of the intervention on overall well-being and life satisfaction.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Çankırı Karatekin University, Çankırı
  - Çakü, Çankırı

IPD SHARING:
Plan to Share IPD: No